CLINICAL TRIAL: NCT05921279
Title: Understanding CARdiac Events in Breast Cancer - Pilot Cardio-Oncology Assessment and Surveillance Pathway for Breast Cancer Patients
Brief Title: Understanding CARdiac Events in Breast Cancer
Acronym: UCARE
Status: Recruiting | Type: Observational
Sponsor: National University of Ireland, Galway, Ireland (Other)
Collaborators: HRB Clinical Research Facility Galway (Other); CORRIB Research Centre for Advanced Imaging and Core Lab, Galway, Ireland (Unknown)
Responsible Party: Principal Investigator, Professor Osama SOLIMAN, Professor of Cardiovascular Research, National University of Ireland, Galway, Ireland
Other Study IDs: C.A. 2890
Record Dates: First submitted 2023-06-19; First posted 2023-06-27 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Breast Cancer; Cardiotoxicity; Cardiomyopathies; Chemotherapeutic Toxicity; Heart Failure; Oncology
Keywords: Cardio oncology
MeSH Terms: conditions — Breast Neoplasms; Cardiotoxicity; Cardiomyopathies; Heart Failure; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bloods for Biobank specimens - Serum, whole blood, paxgene, plasma and serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (4):
- Anthracycline based chemotehrapy low and moderate risk: Patients recieving anthracycline based chemotherapy who fall into the low and moderate risk category following HFA - ICOS cardiac risk assessment as per the European Society of Cardiology Guidelines.
  These patients are monitored taking biobank bloods, bloods, ecg and cardiac echo as per the European Society of Cardiology guidelines whilst receiving chemotherapy.
- Anthracycline based chemotherapy - high and very high risk: Patients who recieving anthracycline who fall into the high and very high risk category following HFA - ICOS cardiac risk assessment as per the European Society of Cardiology Guidelines.
  These patients are monitored taking biobank bloods, bloods, ecg and cardiac echo as per the European Society of Cardiology guidelines whilst receiving chemotherapy.
- Herceptin targeted therapy - low and moderate risk: Patients who are recieving herceptin that fall into the low and moderate risk category following HFA-ICOS cardiac risk assessment as per the European Society of Cardiology Guidelines. These patients are monitored taking biobank bloods, bloods, ecg and cardiac echo as per the European Society of Cardiology Guidelines.
- Herceptin targeted therapy - high and very high risk: Patients who are recieving herceptin that fall into the high and very high risk category following HFA-ICOS cardiac risk assessment as per the European Society of Cardiology Guidelines. These patients are monitored taking biobank bloods, bloods, ecg and cardiac echo as per the European Society of Cardiology Guidelines.

SUMMARY:
In Ireland, over 3,000 patients are diagnosed with breast cancer annually, and 1 in 9 Irish women will be diagnosed with breast cancer in their lifetime. There is evidence that female breast cancer survivors are more likely to die of cardiovascular disease than their age-matched counterparts.

This research is focused on evaluating pathways for identifying, managing, and overcoming side effects of cancer therapies that can negatively impact quality-of-life and overall outcomes for women during and after cancer treatment. The Cardio-oncology research team at GUH plan to capitalize on their expertise in both cancer care and cardiology to develop a care pathway for cancer patients who are at increased risk of developing heart disease.

DETAILED DESCRIPTION:
Establishment of a Cardio-Oncology assessment and surveillance pathway for breast cancer patients undergoing adjuvant systemic chemotherapy at GUH and the assessment of the feasibility of trialing this approach for risk assessment and early detection of CTRCD in a multicenter, prospective RCT which will inform future development of clinical services for cancer patients nationally and later internationally.

Study Design:

This study is a prospective, single arm, pilot feasibility study.

Study Population:

The study will focus on adult female patients diagnosed with stage I-III breast cancer (BC).

Data Analysis and Statistics:

The PCORE Investigators have established collaboration with biostatisticians at the INSIGHT SFI centre for data analytics within University of Galway for analysis of the multi-component dataset from UCARE. Questionnaire data to assess health related QoL (quality of life) and physical activity will be collected at baseline and at 6-monthly intervals at 3, 6 and 12 months throughout the study period. Clinically important differences in physical activity levels or HR-QoL scores will be recorded as per the tool specific scoring systems. Multivariate analysis will be performed for association between HRQoL measures and predictors in patients undergoing breast cancer treatment. Baseline to 6, 12, 18 and 24 month changes in HRQoL over time will be described in subgroups defined by their treatment characteristics and tumor and host response to therapy (both oncologic and cardio-toxic).

ELIGIBILITY:
Inclusion Criteria:

* Women aged ≥ 18 years
* Ability to read and understand English
* Breast Cancer Stage I- III planned to receive systemic chemotherapy

Exclusion Criteria:

* Patients not for systemic chemotherapy with curative intent
* Patients who are unable to co-operate with the study protocol
* Patients who are unable to give informed consent

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Study Population: Adult female patients diagnosed with stage I-III breast cancer receiving chemotherapy.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-01-14 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
The number of participants with successful application of guideline-directed Cardio-Oncology assessments and surveillance. | 2 years
  To calculate the percentage of patients who successfully completed all guideline required investigations for baseline assessments, during and post chemotherapy surveillance i.e. Echocardiography, ECG, and Cardiac biomarkers (troponin and BNP).

SECONDARY OUTCOMES:
The number of participants with cardiovascular disease (CVD) among patients with breast cancer prior to commencement of systemic chemotherapy. | Baseline
  To assess the incidence of CVD at baseline
The number of participants with common risk factors for CTRCD among patients with breast cancer prior to commencement of systemic chemotherapy. | Baseline
  Using the HFA-ICOS risk assessment tool
Incidence of CTRCD in Irish breast cancer patients receiving chemotherapy. | 3M, 6M, 9M, 12M, 24M
  To assess the incidence of CTRCD at all post-therapy timepoints./
The number of participants with successful collection and biobanking specimens among patients with breast cancer undergoing systemic chemotherapy. | Baseline, 3M, 6M, 9M, 12M, 24M
  To collect and biobank relavant samples
The number of participants with successful collection of guideline-required imaging data among patients with breast cancer undergoing systemic chemotherapy. | Baseline, 3M, 6M, 9M, 12M, 24M
  Feasibility of collection of guideline-required imaging data, defined as the number of participants with successful collection of guidelines-required clinical data among patients with breast cancer undergoing systemic chemotherapy.
The number of participants with successful collection of guideline-required clinical data among patients with breast cancer undergoing systemic chemotherapy. | Baseline, 3M, 6M, 9M, 12M, 24M
  Feasibility of collection of guideline-required clinical data, defined as the number of participants with successful collection of guidelines-required clinical data among patients with breast cancer undergoing systemic chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Osama Soliman, MBBCh, PhD, Principal Investigator — NUIG; Aoife Lowery, MBBCh, PhD, Principal Investigator — NUIG; Michael Kerin, MD, PhD, Principal Investigator — NUIG; William Wijns, MD, PhD, Principal Investigator — NUIG
Locations (4):
- Ireland (4):
  - Galway University Hospital, Galway
  - Galway Clinic, Galway
  - Mayo University Hospital, Mayo
  - Sligo General Hospital, Sligo

IPD SHARING:
Plan to Share IPD: Undecided